CLINICAL TRIAL: NCT01681329
Title: Improving Outcomes for Adults With Generalized Anxiety Disorder: Combining Cognitive-Behavioral Treatment and Interpretation Modification Training
Brief Title: Cognitive-Behavioral Treatment and Interpretation Modification Training for Adults With Generalized Anxiety Disorder
Acronym: CBT+IMT-GAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Collaborators: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Université du Québec à Trois-Rivières (Other); Université de Sherbrooke (Other); Toronto Metropolitan University (Other); Brown University (Other)
Responsible Party: Principal Investigator, Michel J Dugas, Ph.D., Professor of Psychology, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOP-82771-12-04
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: Cognitive-behavioral therapy; Interpretation modification training; Randomized clinical trial; Adults
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral therapy with interpretation training (Experimental): 14 sessions of cognitive-behavioral therapy combined with computerized interpretation modification training
  Interventions: Behavioral: Cognitive-behavioral therapy; Other: Interpretation training
- Cognitive-behavioral therapy with non-active training (Active Comparator): 14 sessions of cognitive-behavioral therapy combined with computerized non-active training
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Cognitive-behavioral therapy addressing intolerance of uncertainty, positive beliefs about worry, negative problem orientation, and cognitive avoidance
  Other Names: Intolerance of uncertainty treatment
Other: Interpretation training — Computerized interpretation training using Word-Sentence Association Paradigm
  Other Names: Cognitive bias modification for interpretations
  Arms: Cognitive-behavioral therapy with interpretation training

SUMMARY:
Generalized Anxiety Disorder (GAD) is a condition characterized by chronic and excessive worry and anxiety. Our group has developed a cognitive-behavioural treatment (CBT) for GAD that has been tested in four previous clinical trials. The findings show that 60 to 70% of affected individuals attain GAD remission and that 50 to 55% achieve high endstate functioning following the treatment. Although these numbers are encouraging, there remain a considerable proportion of individuals who do not fully benefit from treatment. In our most recent CIHR-funded treatment study, we assessed the impact of information processing on the efficacy of CBT for GAD. Our findings show: a) that the tendency to negatively interpret ambiguous information at pre-treatment was associated with greater GAD symptoms at post-treatment; and b) that patients who were less successful at changing their negative interpretation style were also less responsive to CBT. Given that computerized interpretation modification training has been shown to be effective for decreasing the negative interpretation style of anxious individuals, the goal of the current proposal is to determine whether such training can augment the efficacy of CBT for adults with GAD. A total of 138 individuals with a primary diagnosis of GAD will be randomly allocated to one of two conditions: a) CBT plus interpretation modification training or b) CBT plus non-active training. CBT will consist of 14 weekly sessions, with interpretation modification training (or non-active training) administered prior to each session. Measures of GAD symptoms, psychopathology, cognitive vulnerability, and interpretation style will be administered at pre-, mid-, and post-treatment, as well as at 6- and 12-month follow-ups. The proposed study will provide information about the efficacy, clinical usefulness, and mechanisms of interpretation modification training in combination with CBT.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is characterized by excessive and uncontrollable worry and anxiety. In Canada, the point prevalence of GAD is 3 to 4%, and the personal and social costs of GAD are well documented. Over the past decade, new cognitive-behavioural treatments have been developed for GAD. Our group has also developed a cognitive-behavioural treatment (CBT) protocol for GAD, which focuses on intolerance of uncertainty. There are now four published randomized clinical trials of the treatment, with results suggesting that it is more efficacious than wait-list control, supportive therapy, and applied relaxation. Although these results are encouraging, 30 to 40% of affected individuals do not attain diagnostic remission and 45 to 50% do not achieve high endstate functioning at post-treatment.

In an effort to augment the efficacy of the treatment protocol for GAD, we have recently examined a broad range of demographic and clinical variables that might predict a limited response to treatment. The results of our analyses suggest that a particular type of cognitive bias plays a key role in determining treatment response. Specifically, patients with a particularly negative interpretation style (i.e., the tendency to negatively interpret ambiguous information) have a greater probability of not attaining remission following CBT (they also show less improvement on other indicators of treatment outcome). In addition, change in interpretation style appears to mediate change in GAD symptoms over the course of CBT. Thus, the data suggest that treatment efficacy could be increased by adding training strategies that specifically address negatively biased interpretations of ambiguous information. Recently, a number of experimental investigations have shown that the tendency to negatively interpret ambiguous information can be decreased using computerized interpretation modification training. In fact, the data show that such changes can be maintained over time, can generalize to new situations, and can lead to corresponding changes in GAD symptoms and anxiety proneness. Thus, it appears that computerized interpretation modification training has the potential to increase the efficacy of current CBT protocols by directly targeting and decreasing the tendency to negatively interpret ambiguous information.

The proposed randomized clinical trial addresses the following question: Can computerized interpretation modification training augment the efficacy of CBT for GAD? A total of 138 individuals with a primary diagnosis of GAD will be randomly allocated to one of two conditions: a) CBT plus interpretation modification training (CBT+IMT) or b) CBT plus non-active training (CBT+NA). CBT will consist of 14 weekly 50-minute sessions targeting intolerance of uncertainty via procedures such as problem-solving training and imaginal exposure. Participants randomized to the experimental condition will receive 10 minutes of computerized interpretation modification training prior to each CBT session. In interpretation modification training, respondents learn to endorse benign combinations and reject negative combinations of sentences and words, thus promoting new associative learning. Participants in the control condition will receive 10 minutes of non-active training, in which each sentence is paired with a word that is unrelated to the sentence or a word that is related to a non-threatening (and typically peripheral) aspect of the sentence. Measures of GAD symptoms, psychopathology, cognitive vulnerability, and interpretation style will be administered at pre-, mid-, and post-treatment, as well as at 6- and 12-month follow-ups. The proposed study will provide information about the efficacy, clinical usefulness, and mechanisms of interpretation modification training in combination with CBT. Given previous findings on the key role of negative interpretation style in anxiety, the proposed study has the potential to increase our understanding and ability to treat individuals with GAD.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of GAD
* Willingness to keep medication status stable while participating in the study
* Willingness to undergo randomization

Exclusion Criteria:

* Change in medication type or dose in 12 weeks before study entry
* Use of herbal products known to have CNS effects in the 2 weeks before study entry
* Evidence of suicidal intent
* Evidence of current substance abuse
* Evidence of current or past schizophrenia, bipolar disorder or organic mental disorder
* Current participation in other trials
* Concurrent psychotherapy during treatment phase of trial
* Evidence of anxiety symptoms due to a general medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-09; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in severity of GAD symptoms assessed by structured interview | Post-treatment (14 weeks)
  Clinician's Severity Rating (CSR) scale of Anxiety Disorders Interview Schedule for DSM-IV (ADIS-IV)
Change from baseline in severity of GAD symptoms | Post-treatment (14 weeks)
  Worry and Anxiety Questionnaire (WAQ)
Change from baseline in severity of worry | Post-treatment (14 weeks)
  Penn State Worry Questionnaire (PSWQ)

SECONDARY OUTCOMES:
Change from baseline in somatic anxiety | Post-treatment (14 weeks)
  Beck Anxiety Inventory (BAI)
Change from baseline in depressive symptoms | Post-treatment (14 weeks)
  Beck Depression Inventory, 2nd edition (BDI-II)
Change from baseline in hostile attitudes | Post-treatment (14 weeks)
  Aggression Questionnaire, Hostility subscale (AQ-Host)
Change from baseline in intolerance of uncertainty | Post-treatment (14 weeks)
  Intolerance of Uncertainty Scale (IUS)
Change from baseline in beliefs about worry | Post-treatment (14 weeks)
  Why Worry, 2nd edition (WW-II)
Change from baseline in problem orientation | Post-treatment (14 weeks)
  Negative Problem Orientation Questionnaire (NPOQ)
Change from baseline in cognitive avoidance | Post-treatment (14 weeks)
  Cognitive Avoidance Questionnaire (CAQ)

OTHER OUTCOMES:
Change from baseline in interpretation of scrambled sentences | Post-treatment (14 weeks)
  Scrambled Sentence Task for GAD (SST-GAD)
Change from baseline in interpretation of ambiguous scenarios | Post-treatment (14 weeks)
  Ambiguous/Unambiguous Situations Diary, Extended version (AUSD-Ext)
Change from baseline in interpretation of ambiguous pictures | Post-treatment (14 weeks)
  Affective Picture Rating Task (APRT)

CONTACTS AND LOCATIONS:
Overall Officials: Michel J. Dugas, Ph.D., Principal Investigator — Concordia University, Montreal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Clinique des troubles anxieux, Montreal, Quebec, Canada